CLINICAL TRIAL: NCT00927862
Title: The Clinical Impact of Applying Pharmacogenetic Algorithms to Individualize Dosing of Warfarin in Patients Being Initiated on Oral Anticoagulation
Brief Title: Applying Pharmacogenetic Algorithms to Individualize Dosing of Warfarin
Acronym: Coumagen-II
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 154-001
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-08

CONDITIONS: Thromboembolism
Keywords: warfarin metabolism; CYP2C9; genotyping; VKORC1; anticoagulation; atrial fibrillation; deep vein thrombosis; pulmonary embolism; Patients initiating warfarin for thromboembolic conditions
MeSH Terms: conditions — Thromboembolism; Vitamin K-Dependent Clotting Factors, Combined Deficiency Of, Type 2; Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard IWPC warfarin dosing algorithm (Active Comparator): Standard International Warfarin Pharmacogenetics Consortium (IWPC) warfarin dosing algorithm.
  Interventions: Genetic: IWPC adapted genotype-guided dosing algorithm for warfarin
- Modified IWPC warfarin dosing algorithm (Experimental): Modified International Warfarin Pharmacogenetics Consortium (IWPC) warfarin dosing algorithm
  Interventions: Genetic: Modified IWPC genetic-guided warfarin dosing algorithm
- Historical controls (Other): The parallel, standard-dosing patient control cohort was identified by a query of the electronic medical records database of the 3 participating hospitals for the time interval spanning enrollment of the randomized pharmacogenetic (PG)-guided cohorts (July 2008 through December 2010). Patients ≥18 years old initiating warfarin therapy with a baseline and at least 1 follow-up international normalized prothrombin time ratio (INR) level between days 3-14 were selected. Initial dose selection and therapy modification was at individual Intermountain-credentialed physician/healthcare provider discretion. Standard management is non-PG based.
  Interventions: Other: Standard of care treatment

INTERVENTIONS:
Genetic: IWPC adapted genotype-guided dosing algorithm for warfarin — Within the first or second dose, apply an International Warfarin Pharmacogenetics Consortium (IWPC) adapted genotype-guided dosing algorithm to determine the daily maintenance dose of warfarin, based on clinical factors (age, sex, weight, height, etc.), and VKORC1 and CYP2C9 genotypes, to individualize the initial dosing of warfarin. (IWPC algorithm submitted for publication, 5-08)
  Note that a second comparison will be made between the combined genotype-guided dosing groups (standard and modified IWPC warfarin dosing algorithms) and a historical comparator group.
  Other Names: IWPC=international warfarin pharmacogenetic collaboration
  Arms: Standard IWPC warfarin dosing algorithm
Genetic: Modified IWPC genetic-guided warfarin dosing algorithm — Within the first or second warfarin dose, apply a modified International Warfarin Pharmacogenetics Consortium (IWPC)-adapted genotype-guided dosing algorithm to determine the daily maintenance dose of warfarin. The active comparator algorithm (see above) will be further modified to account for the temporal pharmacodynamics of warfarin metabolism, e.g., by ignoring the CYP2C9 variants for the first 2 days.
  Note that a second comparison will be made between the combined genotype-guided dosing groups (standard and modified IWPC warfarin dosing algorithms) and a historical comparator group.
  Other Names: IWPC=international warfarin pharmacogenetic collaboration
  Arms: Modified IWPC warfarin dosing algorithm
Other: Standard of care treatment — The parallel, standard-dosing patient control cohort was identified by a query of the electronic medical records databases of the 3 participating hospitals for the time interval spanning enrollment of the randomized pharmacogenetic cohorts (July 2008-December 2010). Patients >=18 years of age initiating warfarin therapy with a baseline and at least 1 follow-up INR level between days 3 and 14 were selected. Initial dose selection and therapy modification was at individual Intermountain-credentialed physician/healthcare provider discretion. Standard management is non-PG-based. A standard (fixed) initial maintenance dose of 5 mg/d is generally assumed.
  Arms: Historical controls

SUMMARY:
The purpose of this study is to determine whether DNA analysis improves the efficiency of dosing and safety in patients who are being started on warfarin therapy.Warfarin, a blood thinner (anticoagulant) prescribed to 1-2 million patients in the United States, is a leading cause of drug-related adverse events (e.g., severe bleeding), in large part due to dramatic (20-fold) differences between individuals in dose requirements. At least half of this variability now can be explained by 3 common genetic variants, age, body size, and sex; however, warfarin therapy continues to begin with the same dose in every patient with the correct individual dose determined by trial and error. This study proposes to determine genetic variations the same day from DNA simply obtained by swabbing the inside of the cheek and use this information to determine the proper dose regimen individually in each patient. The aim is to show that the investigators can achieve more rapid, efficient, and safe dosing in up to 500-1000 individuals who are initiating warfarin therapy for various clotting disorders across a large healthcare system in order to demonstrate improved dosing effectiveness, efficiency, and safety with genetic-based dosing, which could lead to a nationwide application resulting in as much as a $1 billion dollar annual benefit in healthcare outcomes.

DETAILED DESCRIPTION:
Study Objectives:

The specific objectives of CoumaGen-II to be tested are:

1. To apply routine pharmacogenetic (PG)-guided dosing of warfarin in clinical practice at Intermountain Healthcare facilities in the Urban Central Region (i.e., Intermountain Medical Center [IMC], LDS Hospital, Alta View Hospital [AVH]), and selected physician offices that are frequent initiators of warfarin) in a major new quality improvement and clinical research initiative.
2. To compare the percentage out-of-range (%OOR) international normalized prothrombin time ratios (INRs) during the first month (and secondarily, 3 months) of warfarin therapy using PG-guided dosing with parallel or historical standard (STD), empiric dosed controls.
3. To compare a modified PG-guided dosing algorithm (modified-International Warfarin Pharmacogenetics Consortium [IWPC]) with a previously generated and validated, multicenter PG-guided algorithm (IWPC).

Study Design:

Qualifying patients being initiated on warfarin therapy with a target INR of 1.5-2.5, 2-3, or 2.5-3.5 will be invited to participate and sign informed consent. Enrolled patients will receive DNA sampling by buccal swab, and samples will be processed and a PG-guided initial dose calculated with a goal of <6 hours (maximum, 24 hours). Dosing and dose adjustments will be managed through the Urban Central Region (IMC/LDSH) anticoagulation management service (AMS). Dose adjustments through day 8 will use a PG-modified algorithm, after which modification will revert to the standard IHC algorithm. AMS pharmacists and study coordinators will ascertain warfarin doses, INRs, dose changes, and adverse events, and record information on case report forms.

Study Duration:

Each patient will participate for approximately 3 months (90 days ± 10 days). The anticipated enrollment period is 24 months or until 1000 patients are enrolled. The length of the enrollment period is subject to revision as it is dependent on the availability of a robust patient pool.

Further study details on dosing algorithm and genotyping methodology may be provided by Intermountain Healthcare Inc.

ELIGIBILITY:
Inclusion Criteria:

* New participants will be those >=18 years old who are appropriate candidates for and being initiated on warfarin therapy with target international normalized prothrombin time ratio (INR) range of either 2-3 or 2.5-3.5 and with intent to be treated for at least 1 month and willing to sign informed consent.
* Those with target INR 2.5-3.5 may be enrolled with dose adjustment for this higher target per Gage et-al. (i.e., 11% increase in dose).
* Dose modification also will be made for amiodarone based on prior, published experience (i.e., 22% decrease in dose).

Exclusion Criteria:

* Those not appropriate for warfarin (e.g., pregnancy) or for pharmacogenetic (PG)-guided dosing for any reason,
* Those having received rifampin within 3 weeks,
* Those with severe co-morbidities (e.g., creatinine > 2.5,hepatic insufficiency, active malignancy, advanced physiological age, noncompliance risk, expected survival <6 months), and
* Physician or patient preference.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2415 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Anderson, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Healthcare Hospitals and Clinics, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Anderson JL, Horne BD, Stevens SM, Woller SC, Samuelson KM, Mansfield JW, Robinson M, Barton S, Brunisholz K, Mower CP, Huntinghouse JA, Rollo JS, Siler D, Bair TL, Knight S, Muhlestein JB, Carlquist JF. A randomized and clinical effectiveness trial comparing two pharmacogenetic algorithms and standard care for individualizing warfarin dosing (CoumaGen-II). Circulation. 2012 Apr 24;125(16):1997-2005. doi: 10.1161/CIRCULATIONAHA.111.070920. Epub 2012 Mar 19. PMID 22431865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Those >= 18 years and being initiated on warfarin therapy with a target international normalized prothrombin time ratio (INR) of 2-3 or 2.5 -3.5 among participating hospitals and outpatient clinics were invited to participate and sign informed consent.
Pre-assignment Details: If after enrollment, pt was found to be not appropriate for warfarin or pharmacogenetic (PG)-guided dosing or physician preference not to have pt participate they were not randomized. Description below and baseline characteristics report combined PG arms because of similarities but outcome measures report combined and individual PG results.
Groups:
- PG Dosing Patients: Patients who were enrolled in CoumaGen-II and thus, received their warfarin dosing by the PG-dosing algorithms were randomized to receive either standard or modified International Warfarin Pharmacogenetics Consortium [IWPC] warfarin dosing. The IWPC derived and published a common algorithm to predict stable maintenance dose based on ~5000 patients across broad geographic and ethnic/racial groups (N Engl J Med 2009;360:753-764). Hence, we based our standard algorithm on the IWPC algorithm with minor modifications to accommodate different INR targets and smoking status, based on supplemental data from Gage et al (Clini Pharmacol Ther 2008;84:326 -331). The modified IWPC algorithm included 2 further modifications: (1) It ignored the CYP2C9 variant status for the first 2 days; and (2) It used a special dose-revision algorithm based on a day 4 (or day 5) INR after 3 (or 4) warfarin doses.
- Parellel/Historical Controls: A parallel, standard-dosing patient control cohort was identified by a query of the electronic medical records databases of the 3 participating hospitals for the time interval spanning enrollment of the randomized pharmacogenetic-guided cohorts (July 2008 through December 2010). Patients >=18 years of age initiating warfarin therapy with a baseline and at least 1 follow-up INR level between days 3 and 14 were selected. Initial dose selection and therapy modification was at individual Intermountain-credentialed physician/healthcare provider discretion. Standard management is non-PG-based. A standard (fixed) initial maintenance dose of 5 mg/d is generally assumed, with loading doses and clinical-factor modifications not specified.
Period: Overall Study
Arm/Group | PG Dosing Patients | Parellel/Historical Controls
Started | 504 | 1911
Completed | 477 (477 patients evaluated in primary analyses and 488 evaluated in secondary analyses.) | 1866
Not Completed | 27 | 45
Not completed — Missing data needed for endpt analyses | 27 | 45

BASELINE CHARACTERISTICS:
Groups:
- PG Dosing Patients: Patients who were enrolled in CoumaGen-II and thus, received their warfarin dosing by the pharmacogenetic (PG)-dosing algorithms (standard or modified IWPC warfarin algorithms)
- Historical Controls: A parallel, clinical effectiveness comparison group that used an algorithm with standard dosing
- Total: Total of all reporting groups
Arm/Group | PG Dosing Patients | Historical Controls | Total
Number analyzed (Participants) | 504 | 1911 | 2415
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 288 | 1214 | 1502
  >=65 years | 216 | 697 | 913
Age Continuous [Mean (Standard Deviation); unit: years] | 61.3 (14.6) | 57.3 (17.5) | 58.0 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268 | 984 | 1252
  Male | 236 | 927 | 1163
Region of Enrollment [Number; unit: participants]
  United States | 504 | 1911 | 2415

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Out of Range (OOR) International Normalized Prothrombin Time Ratio (INRs) in the Standard and Modified Pharmacogenetic Arms.
Description: The percent of out of range (OOR) international normalized prothrombin time ratio (INRs) in the standard and modified pharmacogentic algorithms at 1 month. To account for laboratory INR-measurement error, a 10% margin outside of the target range was allowed in determination of OOR values, ie, INRs <1.8, >3.3 for INR 2.5 target; <2.25, >3.85 for INR 3.0 target. What is reported is the percent of patients with an OOR INR at 1 month.
Time Frame: 1 month (from day 3 to day 30)
Population: Patients >= 18 years of age who have an indication for initiation of warfarin anticoagulation, gave written informed consent, and met other inclusion/exclusion criteria were studied.
Measure: Mean (95% Confidence Interval); unit: percent
Groups:
- Standard IWPC Warfarin Dosing Algorithm: Standard International Warfarin Pharmacogenetics Consortium (IWPC) warfarin dosing algorithm with minor modification
- Modified IWPC Warfarin Dosing Algorithm: Modified International Warfarin Pharmacogenetics Consortium (IWPC) warfarin dosing algorithm with 3 modifications
Arm/Group | Standard IWPC Warfarin Dosing Algorithm | Modified IWPC Warfarin Dosing Algorithm
Number analyzed (Participants) | 245 | 232
percent | 30.6 [27.6 to 33.7] | 31.8 [28.8 to 34.8]
Statistical Analysis 1: Comparison: Standard IWPC Warfarin Dosing Algorithm vs Modified IWPC Warfarin Dosing Algorithm; Comparisons between groups for primary endpoints were made using the unpaired T-test. All consented, randomized patients who were successfully genotyped and received at least one dose of warfarin with at least one post-dose INR were included in efficacy analyses (modified intention to treat [mITT]); Test type: Non-Inferiority or Equivalence — Based on power calculations and feasibility, the minimum recruitment target for the randomized, PG-guided comparison was set at 500 patients. All qualifying parallel control patients were included, anticipated to number ≥1000. For hypothesis 1, the power to exclude inferiority of the modified PG arm vs standard PG arm at a margin (delta) of 5% with 250 patients per group at a 2-sided alpha <0.05 is 87%, assuming a common standard deviation of 0.20; p < 0.05, t-test, 2 sided — Comparisons between groups for primary endpoints were made using the unpaired T-test; Mean Difference (Final Values) = 0.34, Standard Deviation 0.2

2. Secondary Outcome: The Percent of INRs ≥4 or ≤1.5 for the Modified IWPC Warfarin Algorithm and the Standard IWPC Warfarin Algorithm
Description: The percent of INRs ≥4 or ≤1.5 for the pharmacogenetic (modified IWPC warfarin algorithm and the standard IWPC warfarin) algorithms. What is reported is the percent of patients with INRs ≥4 or ≤1.5 at the end of follow-up.
Time Frame: 3 months (baseline to 3 months or to end of warfarin therapy, whichever occurs first)
Population: All consented, randomized patients who were successfully genotyped and received at least 1 dose of warfarin with at least 1 postdose INR.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Standard IWPC Warfarin Dosing Algorithm | Modified IWPC Warfarin Dosing Algorithm
Number analyzed (Participants) | 250 | 238
percent | 15.2 (20.5) | 15.4 (18.2)

3. Secondary Outcome: The Percent of INRs ≥4 or ≤1.5 or SAEs Among the Modified IWPC Warfarin Algorithm and Standard IWPC Warfarin Algorithm.
Description: What is reported is the percent of patients with INRs ≥4 or ≤1.5 or having experienced a serious adverse event (SAE) at the end of follow-up.
Time Frame: 3 months (from baseline to 3 months or end of warfarin therapy, whichever occurs first)
Population: All patients receiving at least 1 dose of warfarin were included in safety analyses until 1 week after the last warfarin dose
Measure: Number; unit: percent
Arm/Group | Standard IWPC Warfarin Dosing Algorithm | Modified IWPC Warfarin Dosing Algorithm
Number analyzed (Participants) | 250 | 238
percent | 53.6 | 59.2

4. Secondary Outcome: The Number of INRs Measured up to 3 Months in the Pharmacogenetic (PG) (Modified and Standard) Algorithms and Parallel Controls.
Description: What is reported is the mean number of INRs measured/drawn among the patients in each arm.
Time Frame: 1-3 months (from baseline to 3 months or end of warfarin therapy, whichever occurs first)
Population: Patients who were enrolled in CoumaGen-II and thus, received their warfarin dosing by the PG-dosing algorithms (standard or modified IWPC warfarin algorithms) were compared to parallel controls
Measure: Mean (Standard Deviation); unit: INRs
Groups:
- PG Dosing Patients: Patients who were enrolled in CoumaGen-II and thus, received their warfarin dosing by the PG-dosing algorithms (standard or modified IWPC warfarin algorithms)
- Parallel Controls: The parallel, standard-dosing patient control cohort was identified by a query of the electronic medical records databases of the 3 participating hospitals for the time interval spanning enrollment of the randomized PG-guided cohorts (July 2008 through December 2010). Patients >=18 years of age initiating warfarin therapy with a baseline and at least 1 follow-up INR level between days 3 and 14 were selected. Initial dose selection and therapy modification was at individual Intermountain-credentialed physician/healthcare provider discretion. Standard management is non-PG-based. A standard (fixed) initial maintenance dose of 5 mg/d is generally assumed, with loading doses and clinical-factor modifications not specified. However,the same standard INR-based dose-modification algorithm developed and promoted by Intermountain is generally recommended.
Arm/Group | PG Dosing Patients | Parallel Controls
Number analyzed (Participants) | 488 | 1866
INRs | 7.70 (3.99) | 7.47 (7.27)

5. Secondary Outcome: Prediction of a Stable Maintenance Dose Among the Pharmacogenetic (PG)-Guided Dosing Algorithms and the Parallel Controls
Description: Prediction of a stable maintenance dose (within 1 mg/day) among the pharmacogenetic (PG)-guided dosing and the parallel control group. For the parallel control group, an empiric starting dose of 5 mg/day was assumed. What is reported is the percent of patients who had their maintenance dose predicted as described above.
Time Frame: 3 months (from baseline to 3 months or until stable dosing is achieved, whichever occurs first)
Population: Patients who were enrolled in CoumaGen-II and thus, received their warfarin dosing by the PG-dosing algorithms (standard or modified IWPC warfarin algorithms) and had a stable maintenance dose that could be determined were compared to parallel controls
Measure: Number; unit: percent
Arm/Group | PG Dosing Patients | Parallel Controls
Number analyzed (Participants) | 444 | 1866
percent | 63.2 | 37.6

6. Primary Outcome: The Percent of Out of Range (OOR) INRs in Pharmacogenetic-guided Patients and Parallel Controls
Description: The percent of out of range (OOR) INRs in the pharmacogenetic (PG)-dosing (standard + modified IWPC warfarin algorithms) and parallel controls. A 10% margin outside of the target INR range was allowed in determination of OOR values, ie, INRs <1.8, >3.3 for INR 2.5 target; <2.25, >3.85 for INR 3.0 target. What is reported is the percent of patients with OOR INRs at 1 month.
Time Frame: 1 month (from day 3 to day 30)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | PG Dosing Patients | Parallel Controls
Number analyzed (Participants) | 477 | 1866
percent | 31.2 [29.2 to 33.5] | 41.5 [39.9 to 43.2]

7. Primary Outcome: The Percent of Time in Therapeutic Range (TTR) for the Standard and Modified Pharmacogenetic Algorithms.
Description: The percent of time in therapeutic INR range for the standard and modified pharmacogenetic algorithms at 1 month. To account for laboratory INR-measurement error, a 10% margin inside of the target range was allowed in determine TTR values, ie, INRs 1.8-3.3 for INR 2.5 target; 2.25-3.85 for INR 3.0 target. What is reported is the percent of TTR for each patient during 1 month.
Time Frame: 1 month (from baseline to day 30)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | Standard IWPC Warfarin Dosing Algorithm | Modified IWPC Warfarin Dosing Algorithm
Number analyzed (Participants) | 245 | 232
percent | 70.2 [67.2 to 73.3] | 67.5 [64.5 to 70.6]

8. Primary Outcome: The Time in Therapeutic Range (TTR) for the Pharmacogenetic-guided Patients and Parallel Controls
Description: The percent of time in therapeutic INR range for the pharmacogenetic (PG)-dosing (standard + modified IWPC warfarin algorithms) guided patients and parallel controls. To account for laboratory INR-measurement error, a 10% margin inside of the target range was allowed in determine TTR values, ie, INRs 1.8-3.3 for INR 2.5 target; 2.25-3.85 for INR 3.0 target. What is reported is the percent of TTR for each patient during 1 month.
Time Frame: 1 month (from baseline to day 30)
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | PG Dosing Patients | Parallel Controls
Number analyzed (Participants) | 477 | 1866
percent | 68.9 [67.2 to 70.6] | 58.4 [56.8 to 60.0]

9. Secondary Outcome: The Percent of INRs ≥4 or ≤1.5 in the Pharmacogenetic (PG)-Guided Dosing Arms and the Parallel Control Arm
Description: What is reported is the percent of patients with an INR ≥4 or ≤1.5 at the end of follow-up.
Time Frame: 3 months (baseline to 3 months or to end of warfarin therapy, whichever occurs first)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | PG Dosing Patients | Parallel Controls
Number analyzed (Participants) | 488 | 1866
percent | 15.3 (19.4) | 27.4 (32.5)

ADVERSE EVENTS:
Time Frame: Patients were included in the SAE safety analyses if they received an INR measurement on Day 4 or 5 and were taking warfarin. Patients were followed until 3 months after warfarin initiation.
Description: Because only those who received an INR measurement on Day 4 or 5 and were taking warfarin were included in the calculation of the serious adverse events, the numbers in each arm are different from what is reported in the participant flow table.
Arm/Group | PG Dosing Patients | Historical Controls
Serious Adverse Events (participants affected / at risk) | 22/487 | 162/1726
Other Adverse Events (participants affected / at risk) | 75/488 | 511/1866
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PG Dosing Patients (N=487) | Historical Controls (N=1726)
adjudicated death, MI, stroke, thromboembolic event, moderate or severe hemorrhage (Cardiac disorders) | 22 | 162
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PG Dosing Patients (N=488) | Historical Controls (N=1866)
INR >=4 or <=1.5 (Blood and lymphatic system disorders) | 75 | 511 — Number of patients who had an average INR >=4 or <=1.5 at the end of follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes